CLINICAL TRIAL: NCT06137040
Title: Timely Administration of IV Magnesium Sulfate in Patients With a Moderate Asthma Exacerbation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16339
Record Dates: First submitted 2023-10-09; First posted 2023-11-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Asthma in Children; Asthma Attack
Keywords: asthma exacerbation; magnesium sulfate; asthma; asthma attack
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Experiment group will receive magnesium sulfate within the first hour with all of the other first line treatments vs. control group will not receive magnesium sulfate within the first hour of treatment.
Who Masked: Participant, Care Provider
Masking Description: Since the study is randomized, the participant and the provider will not know which group the enrolled patient will be in until the patient is randomized to a group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Magnesium Sulfate in the first hour (Experimental): These patients will receive 40-50 mg/kg IV magnesium sulfate within the first hour of treatment alongside all first line asthma exacerbation therapies (ie inhaled beta agonists, IV steroids).
  Interventions: Drug: Magnesium Sulfate within the first hour
- No Magnesium Sulfate (Placebo Comparator): These patients will not receive IV magnesium sulfate within the first hour of treatment but may receive it later if the provider feels it is clinically necessary.
  Interventions: Other: No Magnesium sulfate within the first hour

INTERVENTIONS:
Drug: Magnesium Sulfate within the first hour — The experimental group will receive 40-50 mg/kg of IV magnesium sulfate will be given to the experimental group alongside the first line asthma therapies (ie inhaled beta agonists, IV steroids). This will be given with a 20 mL/kg normal saline bolus (max 1000 mL) to avoid possible hypotension.
  15-19 kg: 750 mg
  20-29 kg: 1000 mg
  30-39 kg: 1500 mg
  >40 kg: 2000 mg
  Other Names: Magnesium within the first hour
  Arms: Magnesium Sulfate in the first hour
Other: No Magnesium sulfate within the first hour — The control group will not receive IV magnesium sulfate within the first hour of treatment.
  Other Names: No magnesium within the first hour
  Arms: No Magnesium Sulfate

SUMMARY:
This study aims to identify whether early administration of magnesium sulfate in moderate asthma exacerbations can potentially avoid admission, decrease length of stay in the emergency department (ED), decrease length of stay (LOS) in the general hospital floor vs pediatric intensive care unit (PICU), and decrease the need for respiratory support.

DETAILED DESCRIPTION:
Patients ages 5-17 presenting to the OU Children's Hospital Emergency Department from October 2023 to July 2024 will be assigned a respiratory score (RS) upon presentation. Those with a RS between 6-9 (moderate exacerbation) will be screened for inclusion. Eligible patient will then be approached for consent. First line asthma therapies including bronchodilators and steroids will not be delayed for the consent process. Patients who consent will be randomized to the control vs. experimental group once consent is obtained.

The study will not be blinded once a patient is randomized to a group, the provider will know whether the patient will receive weight-based IV magnesium within the first hour (experimental group) or receive standard weight-based IV magnesium sulfate per the provider's clinical judgement (placebo group). Magnesium sulfate dosing for the experimental group will be as follows:

15-19 kg: 750 mg

20-29 kg: 1000 mg

30-39 kg: 1500 mg

>40 kg: 2000 mg

Enrolled patients will have their clinical course reviewed and data obtained regarding LOS in ED and hospital stay, need for respiratory support, and or PICU LOS if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5-17 years old
* Presents to the ED with a respiratory score in the "Moderate" range (6
* Parent(s)/Caregiver(s) speak English

Exclusion Criteria:

* Patients with chronic medical conditions including chronic pulmonary disease (other than asthma), cerebral palsy, congenital heart disease, tracheostomy dependent, myasthenia gravis patients
* Patients who are pregnant
* Parent(s)/Caregiver(s) do not speak English

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Length of Stay in Patients who receive IV Magnesium within the first hour (experimental group) vs control group | From initiation of therapy to discharge from the emergency department or admitting unit, up to 1 week
  Evaluating whether timely administration of IV magnesium sulfate in moderate asthma exacerbations can reduce length of stay in the ED, general hospital bed or PICU. The data will also be analyzed to determine if more patients in the experimental group were able to be discharged from the emergency department compared to the control group.

SECONDARY OUTCOMES:
Evaluate the need for respiratory support in patients receiving magnesium sulfate within the first hour (experimental group) vs control group | Time of initiation of therapy to discharge from the hospital, up to 2 weeks
  Evaluating whether timely administration of IV magnesium sulfate in moderate asthma exacerbations can decrease the need for respiratory support including invasive and non-invasive respiratory support devices.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan McKee, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma Children's Hospital, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheuk DK, Chau TC, Lee SL. A meta-analysis on intravenous magnesium sulphate for treating acute asthma. Arch Dis Child. 2005 Jan;90(1):74-7. doi: 10.1136/adc.2004.050005. PMID 15613519
- [Background] Kokotajlo S, Degnan L, Meyers R, Siu A, Robinson C. Use of intravenous magnesium sulfate for the treatment of an acute asthma exacerbation in pediatric patients. J Pediatr Pharmacol Ther. 2014 Apr;19(2):91-7. doi: 10.5863/1551-6776-19.2.91. PMID 25024668
- [Background] Liu X, Yu T, Rower JE, Campbell SC, Sherwin CM, Johnson MD. Optimizing the use of intravenous magnesium sulfate for acute asthma treatment in children. Pediatr Pulmonol. 2016 Dec;51(12):1414-1421. doi: 10.1002/ppul.23482. Epub 2016 May 24. PMID 27218606
- [Background] Shein SL, Farhan O, Morris N, Mahmood N, Alter SJ, Biagini Myers JM, Gunkelman SM, Kercsmar CM, Khurana Hershey GK, Martin LJ, McCoy KS, Ruddy JR, Ross KR. Adjunctive Pharmacotherapies in Children With Asthma Exacerbations Requiring Continuous Albuterol Therapy: Findings From The Ohio Pediatric Asthma Repository. Hosp Pediatr. 2018 Jan 5;8(2):89-95. doi: 10.1542/hpeds.2017-0088. Online ahead of print. PMID 29305409
- [Background] Torres S, Sticco N, Bosch JJ, Iolster T, Siaba A, Rocca Rivarola M, Schnitzler E. Effectiveness of magnesium sulfate as initial treatment of acute severe asthma in children, conducted in a tertiary-level university hospital: a randomized, controlled trial. Arch Argent Pediatr. 2012 Aug;110(4):291-6. doi: 10.5546/aap.2012.eng.291. English, Spanish. PMID 22859321
- [Background] Rowe BH, Bretzlaff JA, Bourdon C, Bota GW, Camargo CA Jr. Magnesium sulfate for treating exacerbations of acute asthma in the emergency department. Cochrane Database Syst Rev. 2000;2000(2):CD001490. doi: 10.1002/14651858.CD001490. PMID 10796650